CLINICAL TRIAL: NCT05312463
Title: Randomized Double-Blind Clinical Trial of Tongjiang Granule in the Treatment of Patients With Overlapping Gastrointestinal Symptoms of Nonerosive Reflux Disease(NERD) and Epigastric Pain Syndrome(EPS)
Brief Title: Assessment on Effects of Tongjiang Granule in Treating Nonerosive Reflux Disease Overlapping Epigastric Pain Syndrome
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other)
Collaborators: First Affiliated Hospital of Heilongjiang Chinese Medicine University (Other); Yueyang Hospital of Integrated Traditional Chinese and Western Medicine (Unknown); Liuzhou Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021XLA117-3
Record Dates: First submitted 2022-03-03; First posted 2022-04-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Gastroesophageal Reflux; Functional Dysphonia
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tongjiang granule group (Experimental): Experiment group: oral administration of Tongjiang granule with warm water after meal for 1 bag each time for three times a day. The medication period was 4 weeks.
  Interventions: Drug: Tongjiang granule
- Tongjiang granule simulant group (Placebo Comparator): Control group:oral administration of Tongjiang granule simulant with warm water after meal for 1 bag each time for three times a day. The medication period was 4 weeks.
  Interventions: Drug: Tongjiang granule simulant

INTERVENTIONS:
Drug: Tongjiang granule — Tongjiang granules, 1 bag / time, 3 times / day.
  Arms: Tongjiang granule group
Drug: Tongjiang granule simulant — Tongjiang granule simulant,1 bag / time, 3 times / day.
  Arms: Tongjiang granule simulant group

SUMMARY:
Overlapping gastrointestinal symptoms of functional gastrointestinal diseases (FGIDs) is an internationally recognized problem in modern medical diagnosis and treatment. Such patients show more physical symptoms and worse quality of life, resulting in a huge economic burden. At present, FGIDs gastrointestinal symptoms overlap, lack of effective and systematic treatment, and the treatment goal is to improve symptoms.The study plans to carry out a multi center and large sample RCT clinical study of Tongjiang granule in the treatment of overlapping gastrointestinal symptoms of non erosive reflux disease(NERD)and epigastric pain syndrome（EPS, so as to provide high-level evidence-based evidence for the treatment of overlapping symptoms of FGIDs and form a diagnosis and treatment scheme that can be popularized.

DETAILED DESCRIPTION:
Overlapping gastrointestinal symptoms of functional gastrointestinal diseases (FGIDs) is an internationally recognized modern medical treatment problem. More than 40.7% of people worldwide suffer from more than one FGIDs.Gastroesophageal reflux disease (GERD) and functional dyspepsia (FD) are common FGIDs. Clinically, the symptom overlap between GERD and FD is very common. Some studies show that 31.32% of FD and 41.15% of FD overlap GERD overlaps with FD, and the presence of FD reduces the response of GERD patients to proton pump inhibitors (PPIs).At present, the pathogenesis of gastrointestinal symptoms overlap in FGIDs is not clear, and there is a lack of effective and systematic treatment. Non erosive reflux disease (NERD) and epigastric pain syndrome (EPS) are common subtypes of GERD and FD. Nerd accounts for about 70% of GERD patients and EPS accounts for more than 50% of FD patients. Long-term use of PPI can lead to many side effects, even dependency. The treatment of traditional Chinese medicine compound has the characteristics of individualized syndrome differentiation and the advantage of "treating different diseases at the same time". It has a significant effect on the overlap of gastrointestinal symptoms in clinic.

ELIGIBILITY:
Inclusion Criteria:

1. It meets the diagnostic criteria of nonerosive reflex disease(NERD)and epigastric pain syndrome(EPS)
2. It meets the diagnostic criteria of liver-stomach depression-heat syndrome of traditional Chinese medicine
3. Age between 18 and 70 years old
4. Patients have informed consent and are willing to receive corresponding treatment

Exclusion Criteria:

1. Patients with active peptic ulcer, gastrointestinal hemorrhage, severe dysplasia of gastric mucosa or suspected malignant change, achalasia or postoperative achalasia
2. There are other organic diseases of the digestive system (such as acute and chronic pancreatitis, cirrhosis, etc.), or systemic diseases that affect the gastrointestinal motility, such as hyperthyroidism, diabetes mellitus over 10 years, chronic renal insufficiency, spirit (the score of SAS and SDS shows severe anxiety or depression), nervous system diseases, etc
3. Patients with severe organ diseases such as heart, liver and kidney (such as ALT, AST more than 2 times of normal value), hematopoietic system diseases and tumors
4. HP infection was positive (bacterial culture, histological examination, urea breath test, rapid urease test and fecal antigen test were positive);
5. People with a history of gastric / abdominal surgery (excluding appendectomy);
6. Pregnant and lactating women;
7. People with a history of allergies to all the test drugs
8. Subjects who are participating in other clinical trials or have participated in other clinical trials within 4 weeks
9. Other situations that reduce the possibility of enrollment or complicate enrollment according to the judgment of the researcher, such as frequent changes in working environment and other situations that are easy to cause loss of follow-up.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2022-03-26 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale（VAS）scores of main symptoms （heartburn, reflux, epigastric pain, epigastric burning sensation） | 10 weeks
  Observe the changes of VAS scores of main symptoms（heartburn, reflux, epigastric pain, epigastric burning sensation） at baseline and after 2, 4 weeks of medication and 2, 4 and 6 weeks of withdrawal，If the score descends, it indicates that the patient's condition has improved.

SECONDARY OUTCOMES:
Visual Analogue Scale（VAS）scores of Atypical symptoms and other symptom scores （chest pain, pharyngeal foreign body sensation, cough, etc） | 10 weeks
  Observe the changes of VAS scores of Atypical symptoms and other symptom scores（chest pain, pharyngeal foreign body sensation, cough, etc） at baseline and after 2, 4 weeks of medication and 2, 4 and 6 weeks of withdrawal,If the score descends, it indicates that the patient's condition has improved.
the MOS item short from health survey (SF-36 scale) | 10 weeks
  Observe the changes of SF-36 scale at baseline and after 2, 4 weeks of medication and 2, 4 and 6 weeks of withdrawal,if the score descends, it indicates that the patient's condition has improved.
Patient-Reported Outcome (Pro scale) | 10 weeks
  Observe the changes of Pro scale at baseline and after 2, 4 weeks of medication and 2, 4 and 6 weeks of withdrawal,if the score descends, it indicates that the patient's condition has improved.
Hospital Anxiety and Depression Scale (HAD) | 10 weeks
  Observe the changes of Hospital Anxiety and Depression Scale (had) at baseline and after 2, 4 weeks of medication and 2, 4 and 6 weeks of withdrawal,if the score descends, it indicates that the patient's condition has improved.
Visceral Sensitivity Scale (VSI) | 10 weeks
  Observe the changes of Visceral Sensitivity Scale (VSI) at baseline and after 2, 4 weeks of medication and 2, 4 and 6 weeks of withdrawal,if the score descends, it indicates that the patient's condition has improved.

CONTACTS AND LOCATIONS:
Locations (1):
- Xiyuan Hospital of China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No